CLINICAL TRIAL: NCT04435002
Title: The Effect of Acupressure on Fatigue in Individuals With Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01.E.16104
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2020-06

CONDITIONS: Acupressure; Fatigue Syndrome, Chronic; Complementary Therapies; Quality of Life; Depression
Keywords: Acupressure; Fatigue Syndrome, Chronic,; Complementary Therapies
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Depression | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): For 9 different points acupressure technique applied to this group for 4 weeks
  Interventions: Other: Acupressure
- Control Group (No Intervention)

INTERVENTIONS:
Other: Acupressure — Acupressure technics applied to (Liv- 4 , Ht-7 Bilateral, Liv-3 Bilateral, Anmian Bilateral, Yin-Tang unilateral ve Sp-6 Bilateral)
  Arms: Intervention Group

SUMMARY:
Chronic fatigue syndrome is a common problem in society. The treatment of this problem is limited. Acupressure is a treatment method that has become widespread and promising in recent years. For this purpose, the effect of acupressure treatment on chronic fatigue syndrome was investigated.

DETAILED DESCRIPTION:
This study aimed to determine the effectiveness of acupressure technique in individuals with chronic symptoms. In our study, individuals participating in the study will be randomized by the physiotherapist who has received the training of acupressure therapy. The study will be done for a total of 10 sessions for 4 weeks. Individuals' fatigue levels will be measured by Fatigue Severity Scale, their quality of life will be measured by Short Form-36 and depression levels by Beck Depression Inventory. Evaluations will be made at the beginning and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 year old
* Not using any medical treatment,
* Not being included in any physiotherapy program in the last 3 months,
* Does not have any systemic disease,
* Spending at least 4 hours at the computer or desk during the work

Exclusion Criteria:

* Fibromyalgia
* Rheumatoid arthritis
* Open Wound
* Skin Failure

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 5 min
  Min Score:9 Max:63 Greater score shows greater fatigue

SECONDARY OUTCOMES:
Beck Depression Inventory | 15 min
Short Form-36 questionnaire | 15 min

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet